CLINICAL TRIAL: NCT00204568
Title: Randomized Phase II Trial of Trofosfamide vs. Adriamycin in Elderly Patients With Previously Untreated Metastatic Soft Tissue Sarcoma
Brief Title: Trofosfamide Versus Adriamycin in Elderly Patients With Soft Tissue Sarcoma (STS)
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University Hospital Schleswig-Holstein (Other)
Collaborators: Arbeitsgemeinschaft fur Internistische Onkologie (Other); German Sarcoma Group (Other); French Sarcoma Group (Other)
Responsible Party: Principal Investigator, J. T. Hartmann, Prof. Dr. med. J. T. Hartmann, University Hospital Schleswig-Holstein
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: jth_001
Record Dates: First submitted 2005-09-13; First posted 2005-09-20 (Estimated); Last update posted 2013-01-08 (Estimated); Status verified 2013-01

CONDITIONS: Sarcoma, Soft Tissue
MeSH Terms: conditions — Sarcoma | interventions — Doxorubicin; trofosfamide

ARMS (2):
- 1 (Active Comparator): Adriamycin mono
  Interventions: Drug: Adriamycin
- 2 (Experimental): Trofosfamide
  Interventions: Drug: Trofosfamide

INTERVENTIONS:
Drug: Adriamycin — 60 mg/m2, d1, W d22
  Arms: 1
Drug: Trofosfamide — 300 mg absolute d1-7, followed by 150 mg absolute continuously
  Arms: 2

SUMMARY:
The goal of this trial is to determine whether oral continuous (metronomic) therapy with trofosfamide results in a similar rate of progression-free time after 6 months as intravenous treatment with adriamycin. In addition, the study is intended to investigate the level of toxicity associated with the two treatment regimens (safety profile).

DETAILED DESCRIPTION:
Group A:Adriamycin (60 mg/m2, d1, qd22) 75 mg/m2 may be applied instead of 60 mg/m2 for patients between 60 and 70 years of age (optional) Group B:Trofosfamide (300 mg absolute p.o. qd over 7 days, then 150 mg p.o. absolute qd continuously) In case of absence of any toxicity during treatment with trofosfamide 150 mg absolute a dose escalation to 200 mg absolute is allowed (optional)

ELIGIBILITY:
Inclusion Criteria:

* Histologically established metastatic (N+ or M1 = stage IV) or non-resectable soft tissue sarcoma·
* Grading II/III (Guillou et al. J Clin Oncol 1997)
* At least 1 measurable tumor parameter according to RECIST criteria
* Evidence of progression or primary manifestation (except osseous metastases and pleural effusion)
* No previous radiation therapy of the only measurable lesion
* No previous chemotherapy for metastatic disease; previous adjuvant chemotherapy is permitted if there was no progression of the disease within a period of 6 months
* Patients aged 60 years and beyond
* Written patient informed consent
* ECOG Status 0-2
* Granulocytes >= 2 x 10**9/l and thrombocytes >= 100 x 10**/l
* Serum creatinine, bilirubin < 1.5 times the upper limit of normal value, albumin > 25 g/l
* No severe comorbidity including psychosis or any previous history of uncontrolled cardiovascular disease
* Normal left-ventricular function by echocardiography or MUGA scan
* No symptomatic CNS metastases
* Willingness to receive regular follow-up examinations

Exclusion Criteria:

* Histological grading of malignancy: G I
* Histology of gastrointestinal stromal tumor, chondrosarcoma, uterine stromal sarcoma, mesothelioma, neuroblastoma, osteosarcoma, Ewing´s sarcoma/PNET, desmoplastic round cell tumor, embryonal rhabdomyosarcoma, alveolar soft tissue sarcoma
* Less than 5 years free of secondary malignancy except adequately treated carcinoma in situ (CIS) of the cervix, the bladder urothelium, basal cell carcinoma, or adenoma of the colon including pTIS, pTIN

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 117 (Estimated)
Dates: Start 2004-08; Primary Completion 2013-10 (Estimated); Study Completion 2013-10 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival after 6 months | after 6 months
  Progression-free survival after 6 months

SECONDARY OUTCOMES:
Grade III/IV toxicity Objective remission rate according to RECIST criteria Overall survival • Quality of life according to EORTC QLQ-30
  Grade III/IV toxicity Objective remission rate according to RECIST criteria Overall survival Quality of life according to EORTC QLQ-30

CONTACTS AND LOCATIONS:
Overall Officials: Joerg T. Hartmann, MD, Principal Investigator — University Medical Center , Comprehensive Cancer Center North, Christian-Albrechts-University
Locations (1):
- University Medical Center , Comprehensive Cancer Center North, Christian-Albrechts-University, Kiel, Germany